CLINICAL TRIAL: NCT00854373
Title: Concomitant Administration of FSH With HCG Improves Oocyte Maturation and Quality Double -Blinded Randomized Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MR-9999
Record Dates: First submitted 2009-03-02; First posted 2009-03-03 (Estimated); Results first posted 2013-08-05 (Estimated); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Infertility
Keywords: Infertility; Pregnancy; in vitro fertilization
MeSH Terms: conditions — Infertility | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Bravelle
  Interventions: Drug: Bravelle(follicle stimulating hormone)
- 2 (Placebo Comparator): Saline
  Interventions: Other: Saline ( placebo)

INTERVENTIONS:
Drug: Bravelle(follicle stimulating hormone) — One dose of 6 amps of Bravelle given at the same time as HCG ovulation trigger.
  Arms: 1
Other: Saline ( placebo) — 1 cc of Normal Saline (placebo) given at the same time as HCG ovulation trigger.
  Arms: 2

SUMMARY:
Marcelle Cedars, M.D., Victor Fujimoto, M.D., Mitch Rosen, M.D., Heather Huddleston, M.D., Paolo Rinaudo, M.D., Anthony Dobson, M.D., and Shehua Shen, M.D. from the UCSF Department of Obstetrics and Gynecology and Reproductive Sciences are conducting a study to learn about ovarian stimulation and oocyte maturation to improve fertilization, embryo quality, implantation and clinical pregnancy rates in patients undergoing in vitro fertilization (IVF). Two hormones, follicle stimulating hormone and human chorionic gonadotropin (FSH/hCG) will be compared to the standard one hormone, hCG, for the ovulation trigger.

Over the past two decades, the success rate of assisted reproductive technology (ART) has dramatically increased. This increase has largely been attributed to improvements in the laboratory conditions and improvements in ovarian stimulation protocols (those medications used to increase the number of eggs maturing each cycle). Less work has been done on different ways to cause the final maturation of the eggs and the release of the egg from the ovary. The investigators propose to change the final injection prior to the egg retrieval (the ovulation trigger) so that it looks more like what happens in a normal menstrual cycle, where two hormones (both luteinizing hormone (LH) and FSH) increase. The investigators want to find out if this will improve egg quality and increase chances for pregnancy.

DETAILED DESCRIPTION:
We observe during (In vitro fertilization) IVF, there are deviations in oocyte morphology and maturity within an individual cohort and that oocyte degeneration, and failed fertilization exist. Regardless, even if fertilization occurs, a large proportion of embryos fail to progress through the pre-implantation stages of development. In order for fertilization and embryo development to occur, the oocyte must mature or develop "competence". FSH may be a fundamental component to the final stages of oocyte maturation. Evidence suggests that with exogenous ovarian stimulation not all follicles achieve equal vascularity, and hence they are exposed to different amounts of FSH. We hypothesize FSH is required, within each follicle, at the time of ovulation trigger for oocyte maturation and prevention of atresia.

The ovarian stimulation prior to IVF attempts to mimic, and yet augment, normal physiology. The stimulation begins with gonadotropins to rescue antral follicles and stimulate growth. Subsequently hCG, which shares 80% homology with LH, is administered to facilitate maturation of the oocyte. However, the ovulatory phase in the normal menstrual cycle encompasses a concomitant LH and FSH prior to ovulation (see figure).

Maturation is a process whereby the oocyte undergoes changes in preparation for fertilization and embryo development. This entails both nuclear and cytoplasmic transformation. Nuclear maturation pertains to the resumption of meiosis to metaphase II (MII). It is well established that the LH surge is intimately involved in this process. Although the mechanism is not completely known, there are several steps. It is thought germinal vesicle breakdown requires a burst of calcium oscillations. During folliculogenesis, nuclear maturation of the oocyte is normally under tonic inhibition by a putative factor, oocyte-meiotic inhibitor (OMI). Some evidence suggests, prior to ovulation, LH inhibits the release of OMI from either the granulosa or theca cells. OMI likely acts as a paracrine factor and increases cAMP production in the granulosa cells (cumulus), which then acts as a messenger to the oocyte to maintain minimal calcium levels. In addition, LH is thought to decrease the gap junction communication between the cumulus and granulosa. Other evidence points to a putative signal that is synthesized by the granulosa cells, called follicular fluid meiotic activating substance. Both elements involved in nuclear maturation involve LH activity. The induction of LH receptors is via FSH. Under physiologic conditions there is a co-existent FSH surge with the LH surge. LH usually rises about 10 fold from baseline and FSH rises roughly 4 fold from baseline. It is possible that the surge of FSH ensures the required amount of LH receptors to complete nuclear maturation.

Cytoplasmic maturation is more difficult to identify. The process entails the synthesis of new proteins and post-translational modifications of existing proteins to allow for calcium activated pathways facilitating fertilization and embryo development. It is known that there is extensive cross-talk between the oocyte and granulosa cells. Few morphogenetic determinants of cytoplasmic maturation have been identified, but this remains an area of intense investigation From a clinical perspective, it is possible that FSH is required in this process of nuclear and/or cytoplasmic maturation, and that a minimal threshold of FSH may be required to maintain the gap junctions for completion of oocyte development. This evidence may be further supported by in-vitro maturation studies that show that FSH has a stimulatory effect on cytoplasmic and nuclear maturation.

Oocyte degeneration (atresia) is observed in 5-15% of the oocytes at the time of, or after, intracytoplasmic sperm injection. The etiology of degeneration has not been determined. The fate of the oocyte is likely determined prior to oocyte retrieval. At the time of retrieval, the apoptotic process in oocytes destined to undergo atresia has probably already been initiated. Under physiologic conditions, the granulosa cells die prior to the oocyte. There is evidence that atretic follicles have a high androgen to estrogen ratio. It is likely an indication of the deteriorating health of the granulosa cells. It is known that FSH has potent anti-apoptotic activity (inhibition of atresia), and the mechanism may be indirect via estradiol production. There is evidence that FSH primed follicles can grow with LH administration, in spite of low FSH levels. However, observations have shown that this process favors large follicles and that in the smaller follicles a critical ratio of FSH activity to LH activity is needed for survival. In support of this theory, others have suggested there is a narrow therapeutic window for LH. If E2 production is not adequate, LH may be detrimental to the follicle. The LH surge might hasten this process, in those follicles with a relative lack of vascularity (and/or lack of maturity), by a massive development of androgens and a relative lack of aromatase activity.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing in vitro fertilization

Exclusion Criteria:

* risk of ovarian hyperstimulation syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2010-04-20 (Actual); Study Completion 2010-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell P Rosen, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF- Mission Bay, San Francisco, California, United States

REFERENCES:
- [Result] Lamb JD, Shen S, McCulloch C, Jalalian L, Cedars MI, Rosen MP. Follicle-stimulating hormone administered at the time of human chorionic gonadotropin trigger improves oocyte developmental competence in in vitro fertilization cycles: a randomized, double-blind, placebo-controlled trial. Fertil Steril. 2011 Apr;95(5):1655-60. doi: 10.1016/j.fertnstert.2011.01.019. PMID 21315341

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women undergoing a long agonist suppression IVF protocol at one U.S. academic center were recruited to participate
Pre-assignment Details: Between June 2007 and March 2010, 232 participants consented for the study. Prior to randomization date, 44 participants were withdrawn from the study for failing to meet randomization criteria {21 cancelled treatment, 15 had elevated estrogen, 8 required a change in clinical treatment plan for which they no longer met eligibility criteria such as needing serrogacy, freezing all eggs or requiring Pre-Gestational Diagnosis}. 188 participants were randomized and included in the final analysis
Groups:
- Bravelle: Bravelle
  Bravelle(follicle stimulating hormone) : One dose of 6 amps of Bravelle given at the same time as HCG ovulation trigger.
- Placebo: Saline
  Saline ( placebo) : 1 cc of Normal Saline (placebo) given at the same time as HCG ovulation trigger.
Period: Overall Study
Arm/Group | Bravelle | Placebo
Started | 95 | 93
Completed | 95 | 93
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bravelle | Placebo | Total
Number analyzed (Participants) | 95 | 93 | 188
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 95 | 93 | 188
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 93 | 188
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 95 | 93 | 188

OUTCOME MEASURES:

1. Primary Outcome: Mean Fertilization Proportion (2PN/Oocytes Collected)
Description: Number of normally fertilized oocytes (2PNs) divided by the total number of oocytes collected (i.e., not just the number of inseminated metaphase II state (MII) oocytes). This accounted for the possibility of both an enhanced oocyte maturation and improved fertilization of the mature oocytes. This also permitted inclusion of both IVF and intracytoplasmic sperm injection (ICSI) cycles in a way that allowed for evaluation of collective fertilization rates (i.e., typically, the denominator in IVF in calculating fertilization rate is all eggs collected, but in ICSI it is calculated using only the number of MII oocytes injected).
Time Frame: 24 hours after IVF or intracytoplasmic sperm injection (ICSI)
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: proportion of oocytes fertilized
Arm/Group | Bravelle | Placebo
Number analyzed (Participants) | 95 | 93
proportion of oocytes fertilized | 0.63 (0.21) | 0.55 (0.21)

2. Secondary Outcome: Mature Oocyte Recovery Rate Percentage
Description: Likelihood of obtaining an oocyte from a single mature-sized follicle on each ovary. Mature follicles are usually 17mm in diameter or greater.
Time Frame: From the ultrasound done on the HCG trigger date, until the oocyte retrieval time which is up to 36 hours after HCG administration
Measure: Number; unit: percentage of follicles with egg
Arm/Group | Bravelle | Placebo
Number analyzed (Participants) | 95 | 93
percentage of follicles with egg | 69.9 | 57.1

3. Secondary Outcome: Clinical Pregnancy Rate Percentage
Description: The percentage of participants that achieve a clinical pregnancy as confirmed by Fetal heart motion by transvaginal ultrasound
Time Frame: 6 weeks after embryo transfer
Measure: Number; unit: percentage of pregnant participants
Arm/Group | Bravelle | Placebo
Number analyzed (Participants) | 95 | 93
percentage of pregnant participants | 56.8 | 46.2

ADVERSE EVENTS:
Time Frame: Adverse Event Data was collected between initial study visit (At Baseline) and final study visit (5 days after the oocyte retrieval procedure had been completed
Description: Study adverse event and/or serious adverse event do not differ from the clinicaltrials.gov definition.
Arm/Group | Bravelle | Placebo
All-Cause Mortality (participants affected / at risk) | 0/95 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/93
Other Adverse Events (participants affected / at risk) | 0/95 | 0/93

LIMITATIONS AND CAVEATS:
This study was powered to detect difference in fertilization instead of pregnancy outcomes, because the number of patients required to detect a 10% absolute difference in pregnancy rates was too large to be completed at our center (n=387 per group).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes